CLINICAL TRIAL: NCT02513329
Title: Effects of Stellate Ganglion Block (SGB) on Vasomotor Symptoms in Women Receiving Anti-Estrogen Therapy for Breast Cancer
Brief Title: Stellate Ganglion Block (SGB) For Women for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Walega, Associate Professor of Anesthesiology; Chief,Section of Pain Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00200390
Record Dates: First submitted 2015-07-20; First posted 2015-07-31 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Hot Flushes; Hot Flashes
Keywords: Breast Cancer; Anti-estrogens; Hot Flushes; Tamoxifen; Aromatase inhibitors; Hot Flashes
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivicaine (Active Comparator): Stellate Ganglion Block injection with 10 mL .5 % bupivacaine.
  Interventions: Drug: Bupivicaine
- Saline (Sham Comparator): Saline injection (.9 normal saline) 5 ml.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivicaine — A computer-generated 1:1 block randomization scheme will be used to assign participants to receive bupivacaine. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card.10 mL .5% bupivicaine will be administered.
  Other Names: Marcaine
  Arms: Bupivicaine
Drug: Saline — A computer-generated 1:1 block randomization scheme will be used to assign participants to receive saline. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card. 5 mL sterile normal saline will be administered.
  Other Names: Sodium chloride solution
  Arms: Saline

SUMMARY:
Vasomotor symptoms (VMS) affect up to 65% of breast cancer survivors and negatively impact their quality of life. The investigators aim to evaluate the benefit of SGB in symptomatic women with breast cancer who are on anti-estrogens and are seeking relief from moderate to very severe VMS that are adversely affecting health and wellbeing. Women with breast cancer on Tamoxifen, aromatase inhibitors (AIs) or Selective Estrogen Receptor Modulators (SERMS) with moderate to very severe VMS will be enrolled as participants in this study.

DETAILED DESCRIPTION:
Hypotheses: The frequency and intensity of subjective and objective VMS will be significantly lower in women randomized to active SGB as compared to sham controls. Mood, memory, cognition, sleep, and quality of life will all be improved in the treatment group as compared to the sham-control group.

Specific Goals and Objectives:

Goal 1: To determine the effect of stellate ganglion blockade (SGB) for reducing subjective and objective VMS in women with breast cancer on tamoxifen, AIs, or SERMs Goal 2: To evaluate the effect of SGB on mood, memory, cognition, sleep and quality of life in women with breast cancer on tamoxifen, AIs, or SERMs.

We aim to conduct a randomized, single-site, sham-control clinical trial of SGB on VMS in 30 women with breast cancer on anti-estrogen therapy (15 per group). The primary entry criterion will be 28 or more moderate to very severe hot flashes per week. VMS will be measured by self-report on a written daily dairy over a 6-month period. Secondary outcomes include changes in mood, sleep, quality of life, and objective hot flashes measured by ambulatory monitoring (skin-conductance temperature monitoring) for 24 hours at baseline, three months and six months. Memory performance with neurocognitive testing will be done at baseline and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. aged 30 to 70 years
2. 28 or more reported moderate-to-very severe hot flashes per week
3. a minimum of two weeks of VMS diary recording prior to SGB
4. current use of tamoxifen, aromatase inhibitors, or SERMs for a breast cancer indication for at last six months
5. willingness to undergo fluoroscopy-guided SGB or sham treatment.
6. Approval of healthcare provider if ≥ 21 for depression and ≥15 for anxiety on the Depression Anxiety and Stress Scale (DASS)
7. Stable use of Selective Serotonin Reuptake Inhibitors (SSRIs), Selective Norepinephrine Reuptake Inhibitors (SNRIs) if applicable

Exclusion Criteria:

1. conditions that preclude SGB or sham intervention (e.g., anatomic abnormalities of the anterior neck or cervical spine; goiter, cardiac/pulmonary compromise; acute illness/infection; coagulopathy or bleeding disorder; allergic reactions/contraindications to a local anesthetic or contrast dye);
2. use of treatments in the past two months that can affect VMS (e.g., use of oral or transdermal Hormone Treatment (HT) or contraceptives, SERMS,
3. conditions or disorders that can affect performance on cognitive tests (e.g., dementia/mild cognitive impairment; stroke; traumatic brain injury; alcohol/substance use; inability to write, speak, or read in English, English as a second language
4. Mini-Mental State Exam (MMSE) ≥ 28
5. conditions that can affect sleep quality (e.g., use of sleep agents; shift work; etc.)

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Walega, MD, MSCI, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Fogel J, Rubin LH, Kilic E, Walega DR, Maki PM. Physiologic vasomotor symptoms are associated with verbal memory dysfunction in breast cancer survivors. Menopause. 2020 Nov;27(11):1209-1219. doi: 10.1097/GME.0000000000001608. PMID 33110036

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivicaine: Stellate Ganglion Block injection with bupivacaine
  Bupivicaine: A computer-generated 1:1 block randomization scheme will be used to assign participants to receive bupivacaine. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card. 10mL of 0.5% bupivicaine will be administered.
- Saline: Saline injection
  Saline: A computer-generated 1:1 block randomization scheme will be used to assign participants to receive saline. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card. 5 mL of sterile normal saline will be administered.
Period: Overall Study
Arm/Group | Bupivicaine | Saline
Started | 20 | 17
Completed (6 months after intervention follow up period) | 15 | 15
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Population: Number of subjects who consented and randomized to treatment.
Groups:
- Bupivicaine: Stellate Ganglion Block injection with bupivacaine
  Bupivicaine: A computer-generated 1:1 block randomization scheme will be used to assign participants to receive bupivacaine. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card.
- Saline: Saline injection
  Saline: A computer-generated 1:1 block randomization scheme will be used to assign participants to receive saline. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card.
- Total: Total of all reporting groups
Arm/Group | Bupivicaine | Saline | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (7.79) | 54.8 (10.99) | 53.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: (kg/m^2)] | 28.0 (4.26) | 32.84 (6.32) | 30.9 (5.15)
Surgical menopause [Count of Participants; unit: Participants] — Number of participants who have undergone a surgical procedure resulting in menopause.
  Participants | 4 | 3 | 7
Post menopausal [Number; unit: count of participants] — Participants who are post menopausal
  count of participants | 16 | 13 | 29
CES D Depressive Symptoms [Mean (Standard Deviation); unit: score on a scale (0 low-60 high)] — CES D is a 20 question survey where each question is scored 0-3 for a possible score of 0 low possibility of depression to 60. A score of 16 on the survey indicates a possibility of depression.
  score on a scale (0 low-60 high) | 13 (10.32) | 13.38 (12.6) | 13.2 (11.5)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: score on a scale (0 good- 21 poor)] — The PSQI is a 7 component survey which is scored on a likert scale of 0 no disfunction to 3 great disfunction. A score of 0-21 is possible. A score of 21 would indicate worst sleep quality.
  score on a scale (0 good- 21 poor) | 14.43 (4.58) | 12.87 (4.56) | 13.75 (4.57)
Functional Assessment of Cancer (FACT-B [Mean (Standard Deviation); unit: score on a scale (0 poor- 123 good)] — The Functional Assessment of Cancer is a 37 item questionnaire scored using a likert scale of 0 (not at all) - to 4 (very much). The score ranges from 0 (poor) to 123 (good).
  score on a scale (0 poor- 123 good) | 98.09 (24.21) | 99.54 (24.22) | 98.71 (24.21)
Vasomotor Symptoms (Hot Flash) [Mean (Standard Deviation); unit: Number of hot flashes/day] — Vasomotor symptoms (hot flashes) number per day as recorded by the participant using a daily diary.
  Number of hot flashes/day | 11.0 (6.19) | 8.78 (3.09) | 10.04 (4.84)
Objective vasomotor symptoms (Hot Flashes) [Mean (Standard Deviation); unit: Number of hot flashes/day] — Objective vasomotor hot flashes per day identified using a monitor attached non-invasively to paticipants skin.
  Number of hot flashes/day | 15.74 (11.22) | 20.02 (10.95) | 17.59 (11.10)
Intensity of hot flashes (diary) [Mean (Standard Deviation); unit: score on a scale (0-100 most intensity)] — Intensity of hot flashes reported by the participant in a daily diary. Scored on a scale of 0- no intensity to 100 greatest intensity.
  score on a scale (0-100 most intensity) | 33.67 (23.7) | 27.38 (11.83) | 30.94 (18.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Night Sweats From Baseline to 6 Months After Intervention.
Description: Change in number of mean night sweats from baseline to 6 months after intervention using a paper diary (subjective measure of frequency). Number is the change from mean baseline number of night sweats to mean 6 months after procedure (number of ns/month)
Time Frame: 6 months after intervention
Population: 3 subjects in the bupivicaine group data was not available, 2 subjects in the saline treatment group data was not available.
Measure: Mean (Full Range); unit: night sweats/month
Arm/Group | Bupivicaine | Saline
Number analyzed (Participants) | 12 | 13
night sweats/month | 5.46 [0 to 117] | 10.09 [0 to 127]

2. Primary Outcome: Change in Number of Hot Flashes From Baseline to 6 Months After Intervention. [Time Frame: 6 Months After Intervention]
Description: Mean change in number of hot flashes from baseline to 6 months after intervention using a paper diary (subjective measure of frequency). Number is the change from mean baseline number of hot flashes to mean 6 months after procedure (number of ns/month)
Time Frame: 6 months after intervention
Population: 2 in the bupivicaine and 1 in the saline group at 6 months did not respond to interview.
Measure: Mean (Full Range); unit: Hot flashes/month
Arm/Group | Bupivicaine | Saline
Number analyzed (Participants) | 13 | 14
Hot flashes/month | 34.3 [6 to 298] | 172.62 [2 to 1887]

3. Primary Outcome: Intensity of Subjective Hot Flashes (HF) at Baseline and 6 Months
Description: Hot flashes intensity from baseline and at 6 months as reported by the subject using paper diary (subjective) measures of intensity (including mild, severe and very severe HF).Intensity scoring = Frequency*Severity = [(frequency of mild*1)+(frequency of moderate*2) + (frequency of severe*3) + (frequency of very severe*4)].
  Mean intensity of hot flashes at baseline and 6 months. Score on a unlimited scale of 0- infinity based on number of hot flashes. A score on the scale where 0 is good higher scores are worse.
Time Frame: 6 months after stellate ganglion block procedure
Population: 10 subjects in the bupivicane group data not obtained and 4 subjects in the saline group not obtained at six months.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bupivicaine | Saline
Number analyzed (Participants) | 20 | 17
score on a scale
  Hot Flash Intensity Baseline: number analyzed (Participants) | 10 | 13
  Hot Flash Intensity Baseline | 411.4 [151 to 1404] | 229.8 [72 to 531]
  Hot Flash Intensity 6 Months: number analyzed (Participants) | 10 | 13
  Hot Flash Intensity 6 Months | 343.3 [11 to 771] | 594.92 [2 to 3774]

4. Secondary Outcome: Survey Score Changes From Baseline to 6 Months After Intervention Using the Epidemiological Studies-Depression(CES-D) Survey.
Description: Baseline score change compared to the 6 month survey score using the Epidemiological Studies-Depression(CES-D) survey. This survey is a 20-item measure that asks to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. CES-D also provides cutoff scores (e.g., 16 or greater) that aid in identifying individuals at risk for clinical depression
Time Frame: 6 months following intervention
Population: 5 subjects in the bupivicaine group and 2 subjects in the saline group data not available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupivicaine | Saline
Number analyzed (Participants) | 15 | 15
Score on a scale | -.14 (1.14) | 1.16 (1.56)

5. Secondary Outcome: Changes From Baseline of Pittsburg Sleep Quality Inventory (PSQI)
Description: Change in Pittsburg Sleep Quality Inventory (PSQI) between baseline and 6 months post intervention. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: 6 month following intervention
Population: 5 subjects in the bupivicaine group and 2 subject in the saline group data was not available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupivicaine | Saline
Number analyzed (Participants) | 15 | 15
Score on a scale | 10.84 (1.14) | 11.92 (1.10)

ADVERSE EVENTS:
Time Frame: 7 days after the first stellate ganglion block.
Description: Adverse events are collected up to 7 days after the stellate ganglion block procedure.
Arm/Group | Bupivicaine | Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT02513329/Prot_SAP_000.pdf